CLINICAL TRIAL: NCT04399798
Title: A proof-of Concept Study of the Use of Janus Kinase 1 and 2 Inhibitor, Baricitinib, in the Treatment of COVID-19-related Pneumonia
Brief Title: Baricitinib for coRona Virus pnEumonia (COVID-19): a THerapeutic Trial
Acronym: BREATH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carlomaurizio Montecucco, Prof, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001185-11
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Proof-of-concept trial with an exploratory single-arm proof of concept Phase IIa study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baricitinib active treatment (Experimental): Baricitinib 4 mg/day
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — 4 mg/day for 7 days
  Other Names: Olumiant

SUMMARY:
The objective of the study is to assess the efficacy and safety of Baricitinib in the treatment of patients with COVID-19 pneumonia.

This will be a proof-of-concept trial with an exploratory single-arm proof of concept Phase IIa study to assess the efficacy and safety profile of Baricitinib in a limited number of patients with severe acute respiratory syndrome (SARS)-CoV-2 pneumonia. If the initial proof of concept phase will lead to favourable results, an open-label, Phase II, randomized controlled trial will be then designed and performed to confirm the results obtained in the proof of concept phase. The proof-of-concept phase guarantees that no safety issues arise on a limited number of patients in the use of a drug new to the current condition being treated.

DETAILED DESCRIPTION:
Baricitinib 4 mg/daily will be prescribed for 7 days to eligible patients showing signs of acute inflammatory response activation. The primary outcome of the study will be the response to treatment. A patient is considered responder in the absence of either moderate to severe oxygenation impairment or death, whichever occurs first, within 8 days from enrolment. The main secondary outcomes will include the responder rate and mortality at 15 days, the quantification of patients experiencing moderate to severe oxygenation impairment, rate of patients admitted to the intensive care unit, length of hospitalization, mortality at 28 days, rate of re-admission, and adverse events. The duration of the study will be 28 days. In the proof of concept phase, 13 patients will be enrolled; if the responders will be at least 4 patients without safety issues, Baricitinib will be considered for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Ability to obtain informed patient consent noting the limitations of existing knowledge regarding Baricitinib's efficacy and the labeled warning and precautions as the proposed use is outside the approved indication, as well as the presence of known risk of being treated with Baricitinib while the subject of an active infection
* informed Consent as documented by signature
* patients with a confirmed SARS-CoV-2 pneumonia
* adult patients aged 18-74 years old
* infiltrates at chest radiography
* c-reactive protein level greater than 10 mg/dl or ferritin level > 900 ug/L
* Lymphocyte count less than 1500/mmc
* > 200 PaO2/FiO2 ≤ 300

Exclusion Criteria:

* patients aged < 18 years old and ≥ 75 years old
* concomitant bacterial infection
* lymphopenia less than 500/mmc
* hemoglobin < 8 g/dl
* absolute neutrophil count < 1 x 109 cells/L
* requiring continuous positive airway pressure (C-PAP) or mechanical ventilation
* sudden clinical deterioration requiring intensive care unit access
* known hypersensitivity or allergy to the study drug
* Creatinine clearance < 30 mL/min; if the creatinine clearance is between 30 and 60 mL/min the dose of Baricitinib should be reduced to 2 mg/daily
* Severe hepatic impairment (no dose adjustment of Baricitinib is required in mild or moderate hepatic impairment)
* Pregnant or breast-feeding
* Active tuberculosis
* Evidence of active hepatitis B (HBV) (HbsAg positive) or with detectable hepatitis C virus (HCV)-RNA, human immunodeficiency virus (HIV)
* Ongoing, acute diagnosis of deep venous thrombosis/pulmonary embolism (DVT/PE)
* Previous diagnosis of DVT/PE

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Response to treatment: absence of moderate to severe oxygenation impairment (Berlin criteria) | 8 days
  A patient is consider responder in the absence of either moderate to severe oxygenation impairment according to Berlin criteria - measured as Partial pressure of oxygen/fraction inspired oxygen (PaO2/FiO2)
Response to treatment: survival | 8 days
  Absence of death within 8 days from enrollment

SECONDARY OUTCOMES:
To quantify the rate of each of: moderate or severe oxygenation impairment within 8 days | 8 days
  Moderate to severe oxygenation impairment according to Berlin criteria (measured as PaO2/FiO2)
To quantify the rate of each of: moderate or severe oxygenation impairment within 15 days | 15 days
  Moderate to severe oxygenation impairment according to Berlin criteria (measured as PaO2/FiO2)
Mortality | 8 days and 15 days
  To quantify mortality within 8 and 15 days
Peripheral capillary oxygen saturation (SpO2) | 8 days; 15 days
  SpO2 will be assessed with the median and 25th-75th percentiles
Partial pressure of oxygen/fraction inspired oxygen (PaO2/FiO2) | 8 days; 15 days
  PaO2/FiO2 will be assessed with the median and 25th-75th percentiles
To assess the rate of patients admitted to the intensive care unit | 8 days; 15 days
  Number of patients over the number of patients enrolled
To measure the length of hospital stay | 8 days; 15 days
  Median number of days and 25th-75th percentiles
28-day mortality | 28 days
  To quantify 28-day mortality
To quantify the rate of re-admission within 28 days | 28 days
  Number of patients readmitted over the number patients enrolled
To quantify the cumulative incidence and severity of adverse events | 28 days
  Number, type, and severity of adverse events
Interleukin (IL)-1; IL-2; IL-10; IL-6; IL-8; IL-17; IL-2 receptor levels; | 15 days
  Serial serum assessments from baseline up to 15 days
TNFalpha; vascular endothelial growth factor (VEGF); interferon gamma (IFNgamma) levels | 15 days
  Serial serum assessments from baseline up to 15 days
Viral load analyses | 15 days
  Serial assessments from baseline up to 15 days for viral load persistence

CONTACTS AND LOCATIONS:
Overall Officials: Carlomaurizio Montecucco, Prof, Principal Investigator — Rheumatology, IRCCS Fondazione Policlinico S. Matteo, Pavia, Italy; Raffaele Bruno, Prof, Study Chair — Infectious Diseases; IRCCS Fondazione Policlinico S. Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson P, Griffin I, Tucker C, Smith D, Oechsle O, Phelan A, Rawling M, Savory E, Stebbing J. Baricitinib as potential treatment for 2019-nCoV acute respiratory disease. Lancet. 2020 Feb 15;395(10223):e30-e31. doi: 10.1016/S0140-6736(20)30304-4. Epub 2020 Feb 4. No abstract available. PMID 32032529
- [Background] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509